CLINICAL TRIAL: NCT05637853
Title: Telemonitored Fast Track Medical Sequencing for Heart Failure With Reduced Ejection Fraction
Acronym: TELE-FASTER
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TELE-FASTER-HF; 2020-02632 202201899-02 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2022-11-25; First posted 2022-12-05 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Home-monitoring; Medical sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFrEF patients (diagnosed within 3 months or hospitalized for worsening of HFrEF) (Experimental): Standardized sequencing of all for main HFrEF drugs: Betablockers, RAASi, SGLT2i, MRA.
  All patients will be started on an SGLT2i (Empagliflozin or Dapagliflozin) and a betablocker (Metoprolol, Bisoprolol or Carvedilol) right after study inclusion. In the second week, RAASi will be introduced with either angiotensin converting enzyme inhibitor (ACEi)(Ramipril or Enalapril) or angiotensin receptor neprilisyn inhibitor (ARNI)(Sacubitril/Valsartan). If the patient is intolerant to either of these, an angiotensin receptor blocker (ARB)(Candesartan, Losartan, Valsartan) will be introduced. During the following weeks, both BB and ACEi/ARNI/ARB will be up titrated every second week according to the sequencing algoritm. MRA (Spironolactone, Eplerenone) will be introduced and up titrated in week 3 and 7 respectively. If the patient is already on either BB or ACEi/ARNI/ARB/MRA they will continue with the previous prescription and dose until the titration scheme indicates uptitration.
  Interventions: Drug: GDMT

INTERVENTIONS:
Drug: GDMT — Predifined fast uptitration of GDMT for HFrEF with support of home monitoring.

SUMMARY:
Research hypothesis:

Fast telemonitored medical sequencing in patients with heart failure with reduced ejection fraction (HFrEF) is safe and feasible.

Background:

Modern therapy for HFrEF offers a highly effective arsenal of drugs, devices and interventional therapies, yet mortality and morbidity remain high in the cohort. One major problem is that drug therapy introduction and up titration has been very hard to implement in a majority of HFrEF patients. Most previous telemonitoring studies have focused on the continuous monitoring of patients and the monitoring itself has been the main intervention. A potentially more effective way to use telemonitoring in heart failure patients may be to combine the technique with a medical intervention when the patients are most vulnerable to heart failure events. The best therapeutic window lies in the period after newly diagnosed heart failure or right after a recent hospitalization following worsened chronic HFrEF.

Method:

We aim to use telemonitoring for fast sequencing of heart failure drugs for patients with HFrEF.

DETAILED DESCRIPTION:
Our hospital and other centra in "Västra Götalandsregionen" has been exploring telemonitoring in a pilot study that started in 2019 and included 100 patients. This study has used an application from Telia called Telia Health Monitoring (THM). Through this application patients may report both objective parameters such as weight, pulse, blood pressure as well as subjective information for example estimation of symptoms and well-being. Overall, this pilot study has reported good safety data and patient satisfaction. In the present study, we intend to use the same application and health care infrastructure as in the pilot study.

Study synopsis

1. Primary aim:

   The primary aim is to assess effectivness and safety/feasibility of fast telemonitored sequencing of heart failure medications in HFrEF patients.
2. Study population:

   Patients (inpatient or outpatient) with confirmed HFrEF who are either newly diagnosed (within 3 month) or hospitalized for worsening heart failure (within 1 month) and in need of medical sequencing are eligible. Different hospitals within "Västra Götalandsregionen" will participate. Participating centres are Sahlgrenska University hospital/Sahlgrenska, Sahlgrenska University hospital/Östra and Skaraborg Hospital Skövde. The aim is also to recruit Södra Älvsborgs hospital as a centre since all these clinics except for Sahlgrenska University hospital/Sahlgrenska have previous experience of the home monitoring equipment.

   A controll group with HFrEF under standard of care will be retrospecively collected and matched with the intervention group for comparison.
3. Objectives:

   i. Primary objective

   To study safety and feasability of fast telemonitored sequencing in HFrEF patients.

   ii. Secondary objectives

   To investigate whether titration to full target doses or OMT of all four classes of HFrEF medications is achievable within 8 weeks of telemonitored sequencing.

   To investigate the proportion of patients still on full target dosage or OMT after 6 months, 1-, 3- and 5-years follow-up.

   To study levels of N-terminal pro brain natriuretic peptides (NT-proBNP) and other laboratory parameters during fast sequencing of heart failure drugs.

   To investigate if objective signs are observed from telemonitored values in patients non-compliant to the fast titration scheme.

   In depth analyses of reported vital signs and their relation to prescription interruption.

   In depth analyses of health assessment questionnaires evaluating patients experiences of home monitoring.

   Prediction models to identify patients tolerating rapid HF medication titration.

   In depth analyses of health assessment questionnaires evaluating the patients experiences of home monitoring.
4. Study design:

   This is an interventional prospective study. All HFrEF patients eligible for study inclusion will be asked to participate in the telemonitored fast medical sequencing intervention. Patients who do not wish to be included in the intervention arm are going to be followed and titrated according to standard of care, in line with local heart failure treatment guidelines. This approach involves visits to the heart failure outpatient clinic with gradual titration of HFrEF medication.
5. Method:

   The study population in TELE-FASTER-HF is patients with newly diagnosed HFrEF (within three months) or patients who are hospitalized for worsening heart failure (within 1 month) and in need of titration of HFrEF medications. The patients will be screened for eligibility for the study at a first nurse visit at the heart failure out-patient clinic or before discharge from the hospital. Eligible patients need to have access to a smartphone and internet connection at home. Patients are going to be equipped with a telemonitoring equipment. The application from Telia also holds a health assessment questionnaire that can be sent to the out-patient clinic. Blood pressure, pulse and weight are reported daily to a designated heart failure nurse. Every week the patient will be automatically asked to answer the health assessment questionnaire which will be sent to the clinic. All parameters will have specified cut-off values for alerting the designated nurse to take action if needed following standard clinical procedures used by the heart failure nurses. Blood samples will be collected at screening visit and during several steps of medical sequencing in accordance with standard procedures. The purpose is to achieve full titration of all four classes of HFrEF medication within 8 weeks after newly diagnosed heart failure or acute decompensation of chronic heart failure. Each patient will be home monitored for a period of 6 mounts.
6. Medical sequencing:

Sequencing will be initiated and carried out in a standardized format for all patients included in the intervention arm. All patients will be started on an SGLT2i and a betablocker right after study inclusion. In the second week, RAASi will be introduced with either angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor neprilisyn inhibitor (ARNI). If the patient is intolerant to either of these, an angiotensin receptor blocker (ARB) will be introduced. During the following weeks, both BB and ACEi/ARNI/ARB will be up titrated every second week according to the sequencing algoritm, figure 2. MRA will be introduced and up titrated in week 3 and 7 respectively. If the patient is already on either BB or ACEi/ARNI/ARB/MRA they will continue with the previous prescription and dose until the titration scheme indicates up titration.

Eligibility criteria

1. Inclusion criteria:

   Patients diagnosed with HFrEF and without contraindications for either of the following drug classes: SGLT2i, BB, RAASi and MRA.
2. Exclusion criteria:

Estimated glomerular filtration rate (eGFR)<45 ml/min Patients with HFrEF already on treatment with either BB or ACEi/ARNI/ARB and up titrated to >50% of maximal recommended dose.

Patients who do not have access to a smartphone or internet connection at home. Patients not able to comprehend the technical aspects of home monitoring or unable to give informed consent.

Endpoints:

Primary endpoint

Safety and feasibility of fast telemonitored sequencing of heart failure medications in HFrEF patients.

Predefined safety endpoint: incidence of treatment-emergent adverse events up to 180 days from start of sequencing. Changes in vital signs compared to base-line will be recorded. Clinical decision will be based on ESC guidelines for heart failure 2021.

Secondary endpoints:

1. Proportion of patients reaching target doses or OMT of BB, SGLT2i, RAASi and MRA within 8 weeks of medical sequencing with home monitoring.
2. Time to reached target doses or OMT of BB, SGLT2i, RAASi and MRA.
3. Proportion of patients capable of reaching full doses of BB, SGLT2i, RAASi and MRA compared to reported prescriptions from Riks-Svikt.
4. Proportion of patients still on OMT after 1-, 3- and 5-years follow-up compared to prescription patterns from Riks-Svikt.
5. Changes in levels of NTproBNP during home monitored sequencing

Statistical considerations:

The primary aim of this study is to evaluate the feasiblity of predifined fast uptitration of guideline directed heart failure medication with support of home monitoring. No formal power calculation was performed.

Patients with home monitoring will be compared with a control group from Riks-Svikt during long-term follow-up. The patients will be matched for age, gender and heart failure diagnose with controls under standard of care at one year follow-up.

All analyses will be performed with the statistical software R (R v3.5.2; R Foundation for Statistical Computing, Vienna, Austria). Nominal significance levels will be 0.05 and all test performed will be two-sided, when appropriate. All confidence intervals will be 95%. Safety and feasibility endpoints will mainly be presented with descriptive statistics. For descriptive baseline characteristics, categorical data are presented as numbers and percentages and continuous data as means with standard deviation or medians with interquartile range. Cox proportional hazard models will be used to calculate the differences between intervention and control groups in reaching full target dosage or OMT, yielding hazard ratios (HR) with 95% CI.

The initial statistical plan have been re-evaluated and updated on ClinicalTrials.gov on 10th of April 2025.

Ethical consideration:

The study will be conducted in compliance with the ICH Good Clinical Practice Guidelines and in accordance with the ethical principles of the Declaration of Helsinki.

The investigators will ensure that all participants will be given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the study and ensure that all subjects are notified that they are free to discontinue with the study at any time. Signed and dated informed consent will be obtained before conducting any study specific procedure and stored in the Study Master File. A copy of the signed Informed Consent Form will also be given to each participant.

Scientific importance:

The scientific evidence regarding modern heart failure treatment is substantial and there is no doubt regarding these drugs powerful potential in reducing morbidity and improving prognosis in patients with HFrEF. This group of patients is large and the number of patients in need for treatment is increasing. Even so, a large proportion of these patients are not prescribed these drugs and if they are, they do not reach target doses in reasonable time. In fact, a majority of HFrEF patients never reach target doses of heart failure drugs.

This study addresses several unexplored parts of heart failure drug therapy introduction and sequencing. Since there are no previous studies addressing implementation of the latest guidelines for HFrEF drugs using home monitoring, this study has the potential of filling an important scientific gap as well as making a large impact in streamlining therapy for these patients.

Risk/benefit assessment:

This is not an experimental drug intervention. All the drugs used in treatment for HFrEF have been safely used in up titration in several previous studies. The concept of home monitoring in heart failure has been used in previous different trials and has shown to be safe. The patients will be remotely monitored daily by heart failure nurses, in this manner patients will be observed more often than in clinical routine which one could argue even may increases the safety for patients when prescribing heart failure drugs. Furthermore, patients will also be followed by blood sampling repeatedly to avoid any adverse drugs events.

Data storage and management:

Study data will be collected using CRFs. The reason for any excluded data or protocol deviations will be documented in the study report. CRF documentation, study documents and other source data will be retained for at least 10 years after finalization of the study.

Information about the patient involved in the current study, the consent date, name of the study must be recorded, saved and stored according to national regulations in the hospitals electronic medical records (Melior).

All patients will receive a unique study code and the study code list will be kept separately from all other data to assure patient confidentiality. Data analyses will be performed on anonymous data set and study results will be presented on a population level with no possibility to identify unique individual. The results will be presented in scientific peer-reviewed journals.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HFrEF and without contraindications for either of the following drug classes: SGLT2i, BB, RAASi and MRA.

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR)<45 ml/min Patients with HFrEF already on treatment with either BB or ACEi/ARNI/ARB and up titrated to >50% of maximal recommended dose.

Patients who do not have access to a smartphone or internet connection at home. Patients not able to comprehend the technical aspects of home monitoring or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-22 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility of fast telemonitored sequencing of heart failure medications in HFrEF patients | 180 days
  Incidence of treatment-emergent adverse events up to 180 days from start of sequencing.

SECONDARY OUTCOMES:
Proportion of patients reaching full doses or OMT of heart failure drugs with home -monitoring | 8 weeks
  Proportion of patients reaching full doses or OMT of BB, SGLT2i, RAASi and MRA within 8 weeks
Proportion of patients still on full target dosage or OMT in future follow-up | 5 years
  Proportion of patients still on OMT after 6 months, 1, 3 and 5 years follow-up compared to prescription patterns from Riks-Svikt
Changes in levels of NTproBNP during home monitored sequencing | 180 days
  Levels of NTproBNP will be measured during home monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Mellberg, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden